CLINICAL TRIAL: NCT00702143
Title: An Open Label, Parallel Group, Multicenter Study, Evaluating the Safety and Imaging Characteristics of 18F-AV-45 in Healthy Volunteers, Patients With Mild Cognitive Impairment (MCI) and Patients With Alzheimer's Disease (AD)
Brief Title: A Phase II Trial of 18F-AV-45 Positron Emission Tomography (PET) Imaging in Healthy Volunteers, Patients With Mild Cognitive Impairment (MCI) and Patients With Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A05
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AD subjects (Experimental)
  Interventions: Drug: florbetapir F 18
- MCI Subjects (Experimental): MCI (mild cognitive impairment)
  Interventions: Drug: florbetapir F 18
- Healthy controls (Experimental)
  Interventions: Drug: florbetapir F 18

INTERVENTIONS:
Drug: florbetapir F 18 — IV injection, 370MBq (10mCi), single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir

SUMMARY:
Evaluate 18F-AV-45 positron emission tomography (PET) imaging for distinguishing healthy control subjects, from subjects with Alzheimer's disease (AD) or Mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria AD:

* Male or female >=50 years of age
* Meet National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS) criteria for probable AD with MMSE score of 10-24

Inclusion Criteria MCI:

* Male or female >=50 years of age
* Have a Clinical Dementia Rating (CDR) of 0.5
* MMSE >24

Normal subjects:

* Male or female >=50 years of age
* MMSE >=29
* Normal on psychometric test battery at screening
* Provide informed consent

Exclusion Criteria:

* Have a history or current diagnosis of other neurologic disease
* Have had or currently have a diagnosis of other neurodegenerative disease
* Have participated in experimental therapy targeted to amyloid plaque

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (15):
- United States (15):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Costa Mesa, California
  - Research Site, New Haven, Connecticut
  - Research Site, Hallandale, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Sunrise, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Albany, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Bennington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- AD Subjects: Probable Alzheimer's Disease (AD) according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association criteria
- Healthy Controls: cognitively normal (healthy) controls
Period: Overall Study
Arm/Group | AD Subjects | MCI Subjects | Healthy Controls
Started | 45 | 60 | 79
Completed | 45 | 60 | 78
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AD Subjects | MCI Subjects | Healthy Controls | Total
Number analyzed (Participants) | 45 | 60 | 79 | 184
Age Continuous [Mean (Standard Deviation); unit: years] | 75.4 (9.21) | 71.7 (10.23) | 69.4 (11.04) | 71.6 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 33 | 45 | 97
  Male | 26 | 27 | 34 | 87
Region of Enrollment [Number; unit: participants]
  United States | 45 | 60 | 79 | 184

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Amyloid Image Assessment
Description: Three readers blinded to all clinical information classified florbetapir-Positron Emission Tomography (PET) images as either positive for amyloid or negative for amyloid. The majority read was the primary efficacy endpoint for the qualitative evaluation.
Time Frame: 50-60 min after injection
Population: One healthy subject received florbetapir F 18 but due to technical difficulties with the scanner was not imaged and is therefore not included in the efficacy population.
Measure: Number; unit: participants
Arm/Group | AD Subjects | MCI Subjects | Healthy Controls
Number analyzed (Participants) | 45 | 60 | 78
participants
  Positive for amyloid | 34 | 23 | 11
  Negative for amyloid | 11 | 37 | 67
Statistical Analysis 1: Comparison: AD Subjects vs MCI Subjects; Fisher exact test comparing the proportion of amyloid positive subjects between clinical diagnosis groups; Test type: Superiority or Other; p = 0.0002, Fisher Exact
Statistical Analysis 2: Comparison: AD Subjects vs Healthy Controls; Fisher exact test comparing the proportion of amyloid positive subjects between clinical diagnosis groups; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: MCI Subjects vs Healthy Controls; Fisher exact test comparing the proportion of amyloid positive subjects between clinical diagnosis groups; Test type: Superiority or Other; p = 0.0014, Fisher Exact

2. Secondary Outcome: Proportion of Positive Florbetapir-PET Scans
Description: Three readers blinded to all clinical information classified florbetapir-PET images as either positive for amyloid or negative for amyloid. The majority read was used to determine the proportion of positive scans across the three groups.
Time Frame: 50-60 min after injection
Population: as for outcome 1
Measure: Number; unit: percentage of amyoid positive scans
Arm/Group | AD Subjects | MCI Subjects | Healthy Controls
Number analyzed (Participants) | 45 | 60 | 78
percentage of amyoid positive scans | 75.6 [60.5 to 87.1] | 38.3 [26.1 to 51.8] | 14.1 [7.3 to 23.8]

3. Primary Outcome: Mean Cortical to Cerebellum SUVR
Description: Standardized Uptake Value ratio (SUVR) is the ratio of tracer uptake in predefined cortical regions, relative to uptake in the whole cerebellum.
Time Frame: 50-60 min after injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | AD Subjects | MCI Subjects | Healthy Controls
Number analyzed (Participants) | 45 | 60 | 78
SUVR | 1.404 (0.2670) | 1.199 (0.2761) | 1.051 (0.1585)
Statistical Analysis 1: Comparison: AD Subjects vs MCI Subjects vs Healthy Controls; Analysis of variance P value testing for an overall difference in the mean cortical SUVR between the clinical diagnostic groups; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: AD Subjects vs MCI Subjects; Analysis of variance contrast P value testing for difference in the mean cortical SUVR; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: AD Subjects vs Healthy Controls; Analysis of variance contrast P value testing for difference in the mean cortical SUVR; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: MCI Subjects vs Healthy Controls; Analysis of variance contrast P value testing for difference in the mean cortical SUVR; Test type: Superiority or Other; p = 0.0003, ANOVA

ADVERSE EVENTS:
Time Frame: AEs were collected up to 7 days after injection. SAEs were collected up to 30 days after injection.
Groups:
- All Subjects: All subjects receiving florbetapir F 18 injection
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 1/184
Other Adverse Events (participants affected / at risk) | 2/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=184)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=184)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days